CLINICAL TRIAL: NCT02001220
Title: LibeRation From MEchanicaL VEntilAtion and ScrEening Frequency Trial: The RELEASE Trial
Brief Title: Screening Frequency Trial to Identify Weaning Candidates
Acronym: RELEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 151113
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Critically Ill
Keywords: screening; invasive ventilation; mechanical ventilation; weaning; spontaneous breathing trials
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Once daily screening (Active Comparator): Patients will undergo assessments to determine readiness to undergo an SBT once daily.
  Interventions: Procedure: Once daily screening
- At least twice daily screening (Experimental): Patients will undergo assessments to determine readiness to undergo an SBT at least twice daily.
  Interventions: Procedure: At least twice daily screening

INTERVENTIONS:
Procedure: Once daily screening — In the 'once daily screening arm', RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily.
  The initial SBT will be 30-120 minutes in duration and may be conducted with any one of the following techniques: T-piece, CPAP < to 5 cm H2 O or PS < 8 cm H2 O with PEEP < 5 - 10 cm H2O. Higher levels of PEEP (8-10 cm H2O) will be permitted (and recorded) to allow for clinician discretion in conducting SBTs in specific patients (e.g., obese, chronic obstructive pulmonary disease) and use of different humidification strategies. Each centre will choose one technique to be used for all patients enrolled at their centre.
  Arms: Once daily screening
Procedure: At least twice daily screening — In the 'at least twice daily' screening arm patients will be screened at a minimum between approximately 6:00-8:00 hours and 13:00-15:00 hours daily. Initial SBT will be conducted in the same manner as once daily screening arm. Subsequent SBTs will be 30-120 minutes in duration and may be conducted with any one of the following techniques: T-piece, CPAP < to 5 cm H2 O or PS < 8 cm H2 O with PEEP < 5 - 10 cm H2O. Higher levels of PEEP (8-10 cm H2O). Higher levels of PEEP (8-10 cm H2O) will be permitted (and recorded) to allow for clinician discretion in conducting SBTs in specific patients (e.g., obese, chronic obstructive pulmonary disease) and use of different humidification strategies. Each centre will be asked to choose one technique to be used for all patients enrolled at their centre.
  Arms: At least twice daily screening

SUMMARY:
During weaning the work of breathing is transferred from the ventilator back to the patient. Approximately 40% of the time on ventilators is spent weaning. Studies support the use of screening protocols and tests of patient's ability to breathe spontaneously (SBTs) to identify weaning candidates. Once daily screening is the current standard of care. With respiratory therapists (RTs) in Canadian intensive care units (ICUs), a significant opportunity exists to screen patients more frequently, conduct more SBTs, and reduce the time spent on ventilators and in the ICU.

The study is seeking to identify the optimal screening frequency to minimize patients' exposure to invasive ventilation. The RELEASE Trial will evaluate a simple a simple construct: more frequent screening will result In earlier identification of weaning candidates, more frequent SBT's, and less time spent on ventilators and in the ICU. More frequent screening is an appealing intervention because it is sensible, low risk, and represents a cost effective use of current resources. This simple intervention holds promise as a strategy that could change clinical practice, enhance the care delivered to critically ill adults, and improve clinically important outcomes.

DETAILED DESCRIPTION:
Eligible patients (< 65 years of age) will be randomly assigned 1:1 to either 'once daily' or 'at least twice daily' screening for weaning readiness.

After randomization, RTs in participating ICUs will be informed of the allocated study arm and bedside nurses will complete a checklist that documents practices related to sedation, analgesia, delirium, and mobilization before each screening period in both study arms. RTs will conduct weaning readiness assessments either 'once daily' or 'at least twice daily' as per group assignment. The checklists, completed by bedside nurses, will merely record current practices in sedation, analgesia and delirium management, and whether patients are being passively or actively mobilized before SBTs.

In the 'once daily screening arm', RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily. If not yet completed, RTs will prompt RNs to complete the 'practices checklist'. In the 'at least twice daily' screening arm patients will be screened at a minimum between approximately 06:00 - 08:00 hours and 13:00 - 15:00 hours daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hours of the scheduled screening period. Additional screening trials in the 'at least twice daily' screening arm will be permitted at the discretion of the clinical team (RTs and physicians). Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted.

In the event of study inclusion before 10:00 am, both study arms will be initiated on the day of randomization. For patients randomized after 10:00 am, only one assessment will be required in both study arms on day one. Similarly, if patients can breathe spontaneously on PS or trigger spontaneous breaths on volume or pressure AC, volume or pressure SIMV ± PS, PRVC, PAV, VS, or APRV before 10:00 am, then the allocated screening protocol can resume. However if, patients can not be returned to a mode that permits spontaneous breaths (PS) or supports triggered breaths (volume or pressure AC, volume or pressure SIMV ± PS, PRVC, PAV, VS, or APRV) until after 10:00 am, screening will be conducted only once daily in both treatment arms on the day of the return and will resume as per treatment allocation thereafter.

To pass the 'readiness to wean screen' and undergo an SBT, all of the following criteria must be met:

1. The patient must be capable of initiating spontaneous breaths on Pressure Support (PS) or triggering breaths on volume or pressure Assist Control (AC), volume or pressure Synchronized Intermittent Mandatory Ventilation (SIMV) ± PS, Pressure Regulated Volume Control (PRVC) or Airway Pressure Release Ventilation (APRV),
2. The ratio of partial pressure of arterial oxygen to the fractional concentration of inspired oxygen (PaO2/FiO2) greater than or equal to 200 mm Hg,
3. Respiratory rate (RR) less than or equal to 35 breaths/min,
4. Positive end-expiratory pressure (PEEP) less than or equal to 10 cm H2O,
5. Heart rate (HR) less than or equal to 140 beats/min,
6. The ratio of respiratory frequency to tidal volume (f/VT) < 105 breaths/min/L during a 2 minute assessment.

ELIGIBILITY:
Inclusion Criteria:

* Receiving invasive mechanical ventilation for ≥ 24 hours.
* Capable of initiating spontaneous breaths on PS or triggering breaths on volume or pressure AC, volume or pressure SIMV ± PS, PRVC, or APRV.
* With an FiO2 ≤ 70%.
* With a PEEP ≤ 12 cm H₂O.
* < 65 years of age

Exclusion Criteria:

* Patients admitted after cardiopulmonary arrest or with brain death or expected brain death.
* Patients who have evidence of myocardial ischemia in the 24 hour period before enrollment.
* Patients who have received continuous invasive mechanical ventilation for ≥ 2 weeks.
* Patients who have a tracheostomy in situ at the time of screening.
* Patients who are receiving sedative infusions for seizures or alcohol withdrawal.
* Patients who require escalating doses of sedative agents.
* Patients who are receiving neuromuscular blockers or who have known quadriplegia, paraplegia, or 4 limb weakness or paralysis preventing active mobilization (e.g. active range of motion, exercises in bed, sitting at edge of bed, transferring from bed to chair, standing, marching in place, ambulating).
* Patients who are moribund (e.g., at imminent risk for death) or who have limitations of treatment (e.g., withdrawal of support, do not reintubate order, however, do not resuscitate orders will be permitted).
* Patients who have profound neurologic deficits (e.g., large intracranial stroke or bleed) or Glasgow Coma Scale (GCS) ≤ 6.
* Patients who are using modes that automate SBT conduct.
* Patients who are currently enrolled in a confounding study that includes a weaning protocol.
* Patients who were previously enrolled in this trial.
* Patients who have already undergone an SBT.
* Patients who have already undergone extubation [planned, unplanned (e.g. self, accidental)] during the same ICU admission.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate our ability to recruit the desired population (1-2 patients, per centre per month, on average) | 2 years

SECONDARY OUTCOMES:
To evaluate clinician compliance with 'once daily' versus 'at least twice daily' screening assessments and the potential for contamination in the 'once daily' arm | 2 years
  In both arms, compliance rates of at least 80% will be considered acceptable in both arms.
  A contamination rate of less than or equal to 10% in the once daily screening arm will be acceptable.
Assess current practices related to sedation, analgesia and delirium management and mobilization before conducting 'once daily' or 'at least twice daily screening' assessments | 2 years
  We expect that these practices will be recorded at least 80% of the time, when feasible. Strategies utilized in < 60% of assessments (leading to the first SBT) in either arm will be considered potentially important.
Identify barriers (clinician and institutional) to recruitment | 2 years
  Descriptive

OTHER OUTCOMES:
Classify trial participants as requiring (i) simple, (ii) difficult or (iii) prolonged weaning using the 'Task Force on Weaning' definitions. | 2 years
  Descriptive
Obtain preliminary estimates of the impact of the alternative screening strategies ('once daily' vs. 'at least twice daily'') on clinically important outcomes | 2 years
  Clinically important outcomes will include time to first Spontaneous Breathing Trial (SBT) and first successful SBT, time to first extubation and successful extubation, total duration of mechanical ventilation, intensive care unit (ICU) and hospital length of stay, ICU and hospital mortality, use of noninvasive ventilation (NIV) following extubation, complications (self-extubation, tracheostomy, reintubation, proportion requiring prolonged mechanical ventilation)] and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Karen EA Burns, MD, FRCPC, Principal Investigator — St. Michael's Hospital and the Li Ka Shing Knowledge Institute
Locations (8):
- Canada (8):
  - St Paul's Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôpital Saint-Luc, Montreal, Quebec
  - Universite de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Burns KEA, Wong JTY, Dodek P, Cook DJ, Lamontagne F, Cohen A, Mehta S, Kho ME, Hebert PC, Aslanian P, Friedrich JO, Brochard L, Rizvi L, Hand L, Meade MO, Amaral AC, Seely AJ; Canadian Critical Care Trials Group. Frequency of Screening for Weaning From Mechanical Ventilation: Two Contemporaneous Proof-of-Principle Randomized Controlled Trials. Crit Care Med. 2019 Jun;47(6):817-825. doi: 10.1097/CCM.0000000000003722. PMID 30920411